CLINICAL TRIAL: NCT05975489
Title: Influence of the Genetic Polymorphisms in the Effect of Caffeine on Fat Oxidation During Exercise
Brief Title: Genetics in the Effect of Caffeine on Fat Oxidation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UFV_genetic_caffeine
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2022-07

CONDITIONS: Genetic Predisposition; Caffeine; Fat Burn
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caffeine 3mg/kg intake (Experimental): A dose of 3 mg/kg of caffeine (Bulk Powders, Essex, United Kingdom) was ingested before the beginning of each test.
  Interventions: Dietary Supplement: Acute caffeine supplementation
- Caffeine 6mg/kg intake (Experimental): A dose of 6 mg/kg of caffeine (Bulk Powders, Essex, United Kingdom) was ingested before the beginning of each test.
  Interventions: Dietary Supplement: Acute caffeine supplementation
- Placebo intake (Placebo Comparator): A dose of 3 mg/kg of placebo (Cellulose, Guinama, Valencia, Spain) was ingested before the beginning of each test.
  Interventions: Dietary Supplement: Acute caffeine supplementation

INTERVENTIONS:
Dietary Supplement: Acute caffeine supplementation — To evaluate the influence of the time of the day (i.e., morning vs evening) on the effect of caffeine on maximal fat oxidation in women

SUMMARY:
Genetic polymorphism on the effect of oral caffeine intake on fat oxidation during exercise has been studied in active and healthy population performing an incremental test on a cycle ergometer with 3-min stages at workloads from 30 to 70% of maximal oxygen uptake (VO2max). Participants performed this test after the ingestion of a) placebo; b) 3 mg/kg of caffeine; c) 6 mg/kg of caffeine. Fat oxidation rate during exercise was measured by indirect calorimetry. The influence of the CYP1A2 c.-163A>C, GSTP c.313A>G and PGC1a polymorphisms was evaluated to determine the effects on fat oxidation during exercise

DETAILED DESCRIPTION:
Caffeine is a natural stimulant with well-recognized sports performance benefits. Aside its performance-enhancing effect, caffeine has the potential of increasing fat utilization during aerobic exercise at submaximal intensities, lowering-down the contribution of carbohydrate as a fuel. This property of caffeine may provoke a glycogen-sparing effect in the skeletal muscle and liver for exercise situations where carbohydrate availability may be a challenge. Additionally, the capacity of caffeine to enhance fat utilization during exercise could be of interest for improving health outcomes as it may increase the rate of change in body composition in exercise programs. Genetic factors like CYP1A2 c.-163A>C, GSTP c.313A>G and PGC1a c.1444G>A and C>T polymorphisms could be associated with the capacity for fat oxidation during exercise. To date, it is unknown if genetics increases fat oxidation and MFO in the same proportion during morning and evening exercise trials in women. For this reason, the aim of the present study was to evaluate the influence of the tCYP1A2, GSTP and PGC1a polymorphisms on the effect of caffeine on fat oxidation and MFO in active and healthy population. The authors hypothesised that genetics would increase fat oxidation and MFO during exercise and this effect would be of similar magnitude at several caffeine doses.

ELIGIBILITY:
Inclusion Criteria:

To be non-smokers. To have low caffeine intake (i.e., < 50 mg of caffeine per day in the previous 2 months) To show no previous history of cardiopulmonary diseases or having suffered musculoskeletal injuries in the previous 6 months.

Exclusion Criteria:

To have VO2max values below 40 ml/kg/min To be sedentary

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Genotype frequency of CYP1A2 polymorphism | Baseline
  Samples shall be obtained by swabbing and scraping of the buccal mucosa by the participant. The c.-163A>C (rs762551) polymorphism will be used.
Genotype frequency of GSTP polymorphism | Baseline
  Samples shall be obtained by swabbing and scraping of the buccal mucosa by the participant. The c.1444G>A (rs8192678) and C>T (rs17650401) polymorphisms will be used.
Genotype frequency of PGC1a polymorphisms | Baseline
  Samples shall be obtained by swabbing and scraping of the buccal mucosa by the participant. The c.313A>G (rs1695) polymorphism will be used.

SECONDARY OUTCOMES:
FATmax | 2-months
  The intensity of exercise that elicits MFO
MFO | 2-months
  Maximal fat oxidation during exercise
RPE | 2-months
  Rate of percevied exertion during exercise
FAT and CHO oxidation | 2-months
  Fat and carbohydrates oxidation

CONTACTS AND LOCATIONS:
Overall Officials: David Varillas Delgado, Principal Investigator — Universidad Francisco de Vitoria, crta Pozuelo-Majadahonda km 1.800 PC 28223, Madrid, Spain
Locations (1):
- Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Varillas-Delgado D, Coso JD, Munoz A, Aguilar-Navarro M, Gutierrez-Hellin J. Influence of the CYP1A2 c.-163 A > C polymorphism in the effect of caffeine on fat oxidation during exercise: a pilot randomized, double-blind, crossover, placebo-controlled trial. Eur J Nutr. 2024 Oct;63(7):2697-2708. doi: 10.1007/s00394-024-03454-3. Epub 2024 Jul 15. PMID 39007997